CLINICAL TRIAL: NCT03775421
Title: Prospective, Multi-center, Single-arm, Open-label Long-term Study Assessing the Safety, Tolerability, and Effectiveness of Macitentan in Fontan-palliated Adult and Adolescent Subjects
Brief Title: An Upcoming Clinical Study to Measure the Safety and Impact of a Drug Called Macitentan in Teenage and Adult Fontan Patients.
Acronym: RUBATO OL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As The RUBATO DB study (NCT03153137) did not show any benefit of treatment with macitentan in Fontan-palliated participants, the sponsor has decided to terminate the RUBATO OL study (NCT03775421). No new safety observations were made.
Sponsor: Actelion (Industry)
Collaborators: Covance (Industry); Henry Ford Health System (Other); Almac Clinical Technologies (Industry); ActiGraph LLC (Other); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055H302; 2018-002821-45 (EudraCT Number)
Record Dates: First submitted 2018-11-21; First posted 2018-12-14 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Disease With Fontan Circulation
Keywords: Congenital Heart Failure; macitentan; Univentricular Heart; Cavopulmonary Anastomosis; Fontan circulation
MeSH Terms: conditions — Univentricular Heart | interventions — macitentan

STUDY DESIGN:
Intervention Model Description: The study is designed as an open-label (OL), single-arm, multicenter long-term trial in which all adolescent (≥ 12 years) and adult male and female subjects who had previously completed in the parent RUBATO DB study (AC-055H301, NCT03153137) will enroll. The primary objective of the study is to assess the long-term safety and tolerability of macitentan. All efficacy endpoints including the ones listed below are considered as exploratory in nature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label treatment period (Experimental): oral administration of 10 mg macitentan once daily
  Interventions: Drug: macitentan 10 mg

INTERVENTIONS:
Drug: macitentan 10 mg — macitentan 10 mg, film-coated tablet, oral use

SUMMARY:
The aim of this open-label (OL) trial is to study the long-term use of macitentan for up to 2 years in Fontan-palliated adult and adolescent patients beyond the 52 weeks of treatment in the parent RUBATO double-blind (DB) study (AC-055H301, NCT03153137). This OL trial studies the long-term effect of macitentan in Fontan-palliated patients as it is not known if the effect of macitentan is sustained beyond 52 weeks (end of the parent RUBATO DB study). In addition, the trial also studies the long-term safety of macitentan as this is also unknown. Furthermore, the opportunity will be given to patients who were on placebo in the parent RUBATO DB study to receive macitentan 10 mg and benefit from a potentially active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent from the subject and/or a legal representative prior to initiation of any study-mandated procedures.
* Subjects who have completed Week 52 of the parent AC-055H301/RUBATO DB study (NCT03153137)
* Women of childbearing potential must:

  1. have a negative serum pregnancy test prior to first intake of OL study drug, and,
  2. agree to perform monthly pregnancy tests up to the end of the safety follow up (S-FU) period, and,
  3. use reliable methods of contraception from enrollment up to at least 30 days after study treatment discontinuation.

Exclusion Criteria:

* Clinical worsening leading to medical interventions including reoperation of Fontan circulation (Fontan take-down) during the enrollment period
* Systolic blood pressure < 90 mmHg (< 85 mmHg for subjects < 18 years old and < 150 cm of height) at rest
* Criteria related to macitentan use
* Any known factor or disease that may interfere with treatment compliance or full participation in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Francis Briand, MD, Study Director — Actelion
Locations (19):
- United States (2):
  - Massachusetts General Hospital Heart Center, Boston, Massachusetts
  - Providence Medical Research Providence Health Care, Spokane, Washington
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Adult Congenital Heart Disease Unit, Chermside
  - Royal Children's Hospital, Parkville
- CHU de Québec Université Laval, Québec, Quebec, Canada
- China (2):
  - Beijing Anzhen Hospital, Beijing
  - Shanghai Children's Medical Center, Shanghai
- Fakultni nemocnice v Motole, Prague, Czechia
- Rigshospitalet Kardiologisk Klinisk, Copenhagen, Denmark
- France (2):
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Cardiologique Du Haut-Lévêque, Pessac
- Auckland City Hospital, Auckland, New Zealand
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Krakowski Szpital Specjalityczny im. Jana Pawla II, Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw
- National Taiwan University Hospital, Taipei, Taiwan
- Queen Elizabeth Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was enrolled twice with 2 different participant IDs but only 111 participants were enrolled in the study.
Groups:
- Macitentan 10 mg: Participants received macitentan 10 milligrams (mg) tablet orally once daily with or without food from Day 1 until the end of the treatment (129 weeks) or till the sponsor decided to stop this study.
Period: Overall Study
Arm/Group | Macitentan 10 mg
Started | 111
Completed | 1
Not Completed | 110
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 3
Not completed — Death | 1
Not completed — Study Terminated by Sponsor | 94

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 87
  More than one race | 0
  Unknown or Not Reported | 0
  Other | 11
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 10
  CANADA | 4
  CHINA | 5
  CZECH REPUBLIC | 16
  DENMARK | 17
  FRANCE | 7
  NEW ZEALAND | 2
  POLAND | 23
  TAIWAN | 6
  UNITED KINGDOM | 3
  UNITED STATES | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Any AE occurring at or after the study treatment start up to 30 days after end of treatment (EOT) (limits included) within the analysis set was considered to be treatment-emergent.
Time Frame: Up to 133 weeks
Population: The RUBATO open-label extension set (OLES) included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 milligrams (mg).
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Participants | 68

2. Primary Outcome: Number of Participants With Treatment-emergent Serious AEs (TESAEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Any SAE occurring at or after the study treatment start up to 30 days after EOT (limits included) within the analysis set was considered to be TESAEs.
Time Frame: Up to 133 weeks
Population: The RUBATO OLES included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Participants | 18

3. Primary Outcome: Number of Participants With TEAEs Leading to Death
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Any AE occurring at or after the study treatment start up to 30 days after EOT (limits included) within the analysis set was considered to be treatment-emergent.
Time Frame: Up to 133 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Participants | 1

4. Primary Outcome: Number of Participants With TEAEs Leading to Premature Discontinuation of Study Treatment
Description: as for outcome 3
Time Frame: Up to 133 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Participants | 2

5. Primary Outcome: Number of Participants With Treatment-emergent Marked Laboratory Abnormalities up to 30 Days After Study Treatment Discontinuation
Description: Number of participants with treatment-emergent marked laboratory abnormalities (Hemoglobin [gram/Liter {g/L}], Platelets [giga/L {10^9 cells/L}], Leukocytes [10^9 cells/L], Lymphocytes [10^9 cells/L], Neutrophils [10^9 cells/L], Prothrombin International Normalized Ratio [PINR;Ratio], Aspartate Aminotransferase [Units/L {U/L}], Bilirubin [micromoles/L {mcmol/L}], Alkaline Phosphatase [U/L], Glomerular Filtration Rate [milliliter/minute/1.73 meter square], Glucose [millimoles/L {mmol/L}], Potassium [mmol/L], Sodium [mmol/L], Triglycerides [mmol/L] were reported. Abnormalities that occurred after study treatment start and up to 30 days after study treatment discontinuation, that were not present at baseline, were treatment-emergent. Marked laboratory abnormalities reported for at least 1 participant were reported in this outcome measure. >=:greater than or equal to; >:greater than; <:less than; ULN: upper limit of normal; L:Low, H:High, LLL:lower/worse than LL, HHH:higher/worse than HH.
Time Frame: Up to 133 weeks
Population: The RUBATO OLES included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 mg. Here, "n" specifies those participants who were analyzed for each specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 111
Participants
  Hemoglobin: LL<100 | 1
  Platelets: LL (< 75): number analyzed (Participants) | 108
  Platelets: LL (< 75) | 3
  Leukocytes: LLL (< 1.9): number analyzed (Participants) | 107
  Leukocytes: LLL (< 1.9) | 2
  Leukocytes: LL (< 3.0): number analyzed (Participants) | 107
  Leukocytes: LL (< 3.0) | 10
  Lymphocytes: HH (> 4.0): number analyzed (Participants) | 106
  Lymphocytes: HH (> 4.0) | 1
  Neutrophils: LL (< 1.5): number analyzed (Participants) | 106
  Neutrophils: LL (< 1.5) | 3
  PINR: HH (>=1.5 ULN): number analyzed (Participants) | 103
  PINR: HH (>=1.5 ULN) | 4
  PINR: HHH (>= 2.5 ULN): number analyzed (Participants) | 103
  PINR: HHH (>= 2.5 ULN) | 1
  Aspartate Aminotransferase: HH (>=3 ULN) | 1
  Bilirubin: HH (>=2 ULN): number analyzed (Participants) | 107
  Bilirubin: HH (>=2 ULN) | 1
  Alkaline Phosphatase: HH (> 2.5 ULN): number analyzed (Participants) | 106
  Alkaline Phosphatase: HH (> 2.5 ULN) | 1
  GFR: LL (< 60): number analyzed (Participants) | 106
  GFR: LL (< 60) | 1
  Glucose: LL (< 3.0): number analyzed (Participants) | 106
  Glucose: LL (< 3.0) | 2
  Glucose: HH (> 8.9): number analyzed (Participants) | 106
  Glucose: HH (> 8.9) | 3
  Potassium: HH (>5.5): number analyzed (Participants) | 106
  Potassium: HH (>5.5) | 1
  Sodium: LLL (<130): number analyzed (Participants) | 106
  Sodium: LLL (<130) | 1
  Triglycerides: HH (>3.42): number analyzed (Participants) | 106
  Triglycerides: HH (>3.42) | 3

6. Primary Outcome: Change From Baseline in Hemoglobin Over Time
Description: Change from baseline in hemoglobin over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: The RUBATO OLES included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 mg. Here, "N" (overall number of participants analyzed) specifies number of participants evaluable for this outcome measure and; "n" specifies those participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 98
g/L
  Week 26 | -6.0 (9.94)
  Week 52: number analyzed (Participants) | 75
  Week 52 | -4.0 (9.19)
  Week 78: number analyzed (Participants) | 42
  Week 78 | -5.0 (7.20)
  Week 104: number analyzed (Participants) | 18
  Week 104 | -2.4 (10.66)
  Week 130: number analyzed (Participants) | 3
  Week 130 | 5.7 (19.35)

7. Primary Outcome: Change From Baseline in Hematocrit Over Time
Description: Change from baseline in hematocrit over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: The RUBATO OLES included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 mg. Here, "N" (number of participants analyzed) specifies number of participants evaluable for this outcome measure and; "n" specifies those participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: Liters/Liter (L/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 100
Liters/Liter (L/L)
  Week 26 | -0.016 (0.0323)
  Week 52: number analyzed (Participants) | 74
  Week 52 | -0.007 (0.0288)
  Week 78: number analyzed (Participants) | 42
  Week 78 | -0.011 (0.0247)
  Week 104: number analyzed (Participants) | 18
  Week 104 | -0.008 (0.0285)
  Week 130: number analyzed (Participants) | 3
  Week 130 | 0.010 (0.0624)

8. Primary Outcome: Change From Baseline in Leukocytes, Neutrophils, Lymphocytes, and Platelets Over Time
Description: Change from baseline in leukocytes, neutrophils, lymphocytes, and platelets over time were reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 100
10^9 cells/L
  Leukocytes: Week 26 | -0.358 (1.2966)
  Leukocytes: Week 52: number analyzed (Participants) | 75
  Leukocytes: Week 52 | -0.222 (1.3677)
  Leukocytes: Week 78: number analyzed (Participants) | 42
  Leukocytes: Week 78 | -0.300 (1.2868)
  Leukocytes: Week 104: number analyzed (Participants) | 18
  Leukocytes: Week 104 | -0.255 (1.2914)
  Leukocytes: Week 130: number analyzed (Participants) | 3
  Leukocytes: Week 130 | -0.560 (1.1186)
  Neutrophils: Week 26: number analyzed (Participants) | 98
  Neutrophils: Week 26 | -0.185 (1.0712)
  Neutrophils: Week 52: number analyzed (Participants) | 75
  Neutrophils: Week 52 | -0.074 (1.0624)
  Neutrophils: Week 78: number analyzed (Participants) | 42
  Neutrophils: Week 78 | -0.233 (1.0569)
  Neutrophils: Week 104: number analyzed (Participants) | 18
  Neutrophils: Week 104 | -0.105 (1.1060)
  Neutrophils: Week 130: number analyzed (Participants) | 3
  Neutrophils: Week 130 | -0.400 (1.0130)
  Lymphocytes: Week 26: number analyzed (Participants) | 98
  Lymphocytes: Week 26 | -0.153 (0.3176)
  Lymphocytes: Week 52: number analyzed (Participants) | 75
  Lymphocytes: Week 52 | -0.098 (0.5366)
  Lymphocytes: Week 78: number analyzed (Participants) | 42
  Lymphocytes: Week 78 | -0.016 (0.3046)
  Lymphocytes: Week 104: number analyzed (Participants) | 18
  Lymphocytes: Week 104 | -0.089 (0.3181)
  Lymphocytes: Week 130: number analyzed (Participants) | 3
  Lymphocytes: Week 130 | -0.113 (0.2223)
  Platelets: Week 26 | -9.2 (24.94)
  Platelets: Week 52: number analyzed (Participants) | 74
  Platelets: Week 52 | -4.3 (30.54)
  Platelets: Week 78: number analyzed (Participants) | 42
  Platelets: Week 78 | -8.1 (24.18)
  Platelets: Week 104: number analyzed (Participants) | 18
  Platelets: Week 104 | -11.1 (25.08)
  Platelets: Week 130: number analyzed (Participants) | 3
  Platelets: Week 130 | 6.7 (12.74)

9. Primary Outcome: Change From Baseline in Systolic and Diastolic Arterial Blood Pressure (BP) Over Time
Description: Change from baseline in systolic and diastolic arterial BP over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 101
millimeters of mercury (mmHg)
  Systolic BP: Week 26 | -0.7 (13.00)
  Systolic BP: Week 52: number analyzed (Participants) | 75
  Systolic BP: Week 52 | -1.7 (14.81)
  Systolic BP: Week 78: number analyzed (Participants) | 43
  Systolic BP: Week 78 | -0.7 (14.79)
  Systolic BP: Week 104: number analyzed (Participants) | 18
  Systolic BP: Week 104 | 0.7 (6.49)
  Systolic BP: Week 130: number analyzed (Participants) | 3
  Systolic BP: Week 130 | -12 (8.72)
  Diastolic BP: Week 26 | -2.9 (12.63)
  Diastolic BP: Week 52: number analyzed (Participants) | 75
  Diastolic BP: Week 52 | -0.9 (12.56)
  Diastolic BP: Week 78: number analyzed (Participants) | 43
  Diastolic BP: Week 78 | -1.6 (11.61)
  Diastolic BP: Week 104: number analyzed (Participants) | 18
  Diastolic BP: Week 104 | 2.6 (9.65)
  Diastolic BP: Week 130: number analyzed (Participants) | 3
  Diastolic BP: Week 130 | -0.7 (7.23)

10. Primary Outcome: Change From Baseline in Pulse Rate Over Time
Description: Change from baseline in pulse rate over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 101
beats per minute (bpm)
  Week 26 | -2.1 (10.48)
  Week 52: number analyzed (Participants) | 75
  Week 52 | 0.9 (10.95)
  Week 78: number analyzed (Participants) | 43
  Week 78 | -1.3 (10.12)
  Week 104: number analyzed (Participants) | 18
  Week 104 | -1.7 (8.78)
  Week 130: number analyzed (Participants) | 3
  Week 130 | -0.3 (13.05)

11. Primary Outcome: Change From Baseline in Peripheral Oxygen Saturation (SpO2) Over Time
Description: Change from baseline in SpO2 over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of SpO2 (%)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 99
percentage of SpO2 (%)
  Week 26 | 0.2 (3.22)
  Week 52: number analyzed (Participants) | 75
  Week 52 | 0.2 (2.79)
  Week 78: number analyzed (Participants) | 43
  Week 78 | -0.5 (2.52)
  Week 104: number analyzed (Participants) | 18
  Week 104 | 0.3 (2.44)
  Week 130: number analyzed (Participants) | 3
  Week 130 | 3.3 (2.31)

12. Primary Outcome: Change From Baseline in Body Weight Over Time
Description: Change from baseline in body weight over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 102
kilograms (kg)
  Week 26 | 0.8 (2.89)
  Week 52: number analyzed (Participants) | 75
  Week 52 | 0.9 (4.23)
  Week 78: number analyzed (Participants) | 43
  Week 78 | 1.7 (3.65)
  Week 104: number analyzed (Participants) | 18
  Week 104 | 2.0 (4.17)
  Week 130: number analyzed (Participants) | 3
  Week 130 | 2.6 (5.54)

13. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (AP), and Gamma Glutamyl Transferase (GGT) Over Time
Description: Change from baseline in ALT, AST, AP, and GGT over time were reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 103
U/L
  ALT: Week 26: number analyzed (Participants) | 101
  ALT: Week 26 | -2.0 (8.57)
  ALT: Week 52: number analyzed (Participants) | 75
  ALT: Week 52 | -2.1 (10.40)
  ALT: Week 78: number analyzed (Participants) | 43
  ALT: Week 78 | -2.7 (11.32)
  ALT: Week 104: number analyzed (Participants) | 18
  ALT: Week 104 | -6.8 (15.72)
  ALT: Week 130: number analyzed (Participants) | 3
  ALT: Week 130 | -13.7 (23.69)
  AST: Week 26: number analyzed (Participants) | 100
  AST: Week 26 | -1.3 (8.39)
  AST: Week 52: number analyzed (Participants) | 75
  AST: Week 52 | -1.7 (9.60)
  AST: Week 78: number analyzed (Participants) | 42
  AST: Week 78 | -3.0 (11.39)
  AST: Week 104: number analyzed (Participants) | 18
  AST: Week 104 | -6.1 (17.03)
  AST: Week 130: number analyzed (Participants) | 3
  AST: Week 130 | -21.3 (41.43)
  AP: Week 26 | -7.7 (36.04)
  AP: Week 52: number analyzed (Participants) | 75
  AP: Week 52 | -1.9 (25.25)
  AP: Week 78: number analyzed (Participants) | 43
  AP: Week 78 | -6.6 (28.02)
  AP: Week 104: number analyzed (Participants) | 18
  AP: Week 104 | -21.8 (53.46)
  AP: Week 130: number analyzed (Participants) | 3
  AP: Week 130 | 6.7 (6.03)
  GGT: Week 26 | -1.2 (14.85)
  GGT: Week 52: number analyzed (Participants) | 75
  GGT: Week 52 | 1.2 (15.74)
  GGT: Week 78: number analyzed (Participants) | 43
  GGT: Week 78 | -2.2 (18.26)
  GGT: Week 104: number analyzed (Participants) | 18
  GGT: Week 104 | -3.2 (18.13)
  GGT: Week 130: number analyzed (Participants) | 3
  GGT: Week 130 | 1.0 (13.23)

14. Primary Outcome: Change From Baseline in Bilirubin, Direct Bilirubin, and Creatinine Over Time
Description: Change from baseline in bilirubin, direct bilirubin, and creatinine over time were reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 103
micromoles per liter (mcmol/L)
  Bilirubin: Week 26 | -0.9 (6.62)
  Bilirubin: Week 52: number analyzed (Participants) | 75
  Bilirubin: Week 52 | -1.1 (10.41)
  Bilirubin: Week 78: number analyzed (Participants) | 43
  Bilirubin: Week 78 | -0.5 (5.68)
  Bilirubin: Week 104: number analyzed (Participants) | 18
  Bilirubin: Week 104 | -0.8 (6.13)
  Bilirubin: Week 130: number analyzed (Participants) | 3
  Bilirubin: Week 130 | -1.3 (2.89)
  Direct Bilirubin: Week 26: number analyzed (Participants) | 101
  Direct Bilirubin: Week 26 | -0.1 (1.14)
  Direct Bilirubin: Week 52: number analyzed (Participants) | 72
  Direct Bilirubin: Week 52 | 0.0 (1.29)
  Direct Bilirubin: Week 78: number analyzed (Participants) | 41
  Direct Bilirubin: Week 78 | 0.0 (1.00)
  Direct Bilirubin: Week 104: number analyzed (Participants) | 18
  Direct Bilirubin: Week 104 | -0.2 (1.25)
  Direct Bilirubin: Week 130: number analyzed (Participants) | 3
  Direct Bilirubin: Week 130 | -1.0 (1.00)
  Creatinine: Week 26: number analyzed (Participants) | 102
  Creatinine: Week 26 | 0.2 (9.27)
  Creatinine: Week 52: number analyzed (Participants) | 75
  Creatinine: Week 52 | 0.9 (9.16)
  Creatinine: Week 78: number analyzed (Participants) | 42
  Creatinine: Week 78 | 0.8 (8.22)
  Creatinine: Week 104: number analyzed (Participants) | 18
  Creatinine: Week 104 | 0.1 (8.10)
  Creatinine: Week 130: number analyzed (Participants) | 3
  Creatinine: Week 130 | -0.7 (5.51)

15. Primary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) Over Time
Description: Change from baseline in GFR over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliters/minute/1.73 meter square
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 102
milliliters/minute/1.73 meter square
  Week 26 | -0.9 (15.43)
  Week 52: number analyzed (Participants) | 75
  Week 52 | -2.0 (15.22)
  Week 78: number analyzed (Participants) | 42
  Week 78 | -0.5 (13.26)
  Week 104: number analyzed (Participants) | 17
  Week 104 | 0.4 (17.00)
  Week 130: number analyzed (Participants) | 3
  Week 130 | -1.7 (7.57)

16. Primary Outcome: Change From Baseline in Prothrombin Time Over Time
Description: Change from baseline in prothrombin time over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 98
seconds
  Week 26 | -0.31 (3.523)
  Week 52: number analyzed (Participants) | 73
  Week 52 | -0.05 (4.038)
  Week 78: number analyzed (Participants) | 42
  Week 78 | -0.38 (2.293)
  Week 104: number analyzed (Participants) | 18
  Week 104 | -1.12 (3.317)
  Week 130: number analyzed (Participants) | 3
  Week 130 | -0.57 (0.651)

17. Primary Outcome: Change From Baseline in Prothrombin International Normalized Ratio Over Time
Description: Change from baseline in prothrombin international normalized ratio over time was reported in this outcome measure.
Time Frame: Baseline up to Week 130
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 98
ratio
  Week 26 | -0.06 (0.401)
  Week 52: number analyzed (Participants) | 73
  Week 52 | -0.06 (0.456)
  Week 78: number analyzed (Participants) | 42
  Week 78 | -0.12 (0.245)
  Week 104: number analyzed (Participants) | 18
  Week 104 | -0.16 (0.379)
  Week 130: number analyzed (Participants) | 3
  Week 130 | -0.07 (0.058)

18. Secondary Outcome: Change From Baseline in Peak Oxygen Uptake/Consumption (VO2)
Description: Change from baseline in peak VO2 was reported in this outcome measure.
Time Frame: Baseline, Week 52, and Week 104
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milliliters per kilogram per minute
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 71
Milliliters per kilogram per minute
  Week 52 | -0.82 (2.724)
  Week 104: number analyzed (Participants) | 12
  Week 104 | -0.93 (1.968)

19. Secondary Outcome: Change From Baseline in Mean Count Per Minute of Daily Physical Activity Measured by Accelerometer (PA-Ac)
Description: Change from baseline in mean count per minute of daily PA-Ac was reported in this outcome measure.
Time Frame: Baseline, Week 26, Week 52, Week 78, and Week 104
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mean count per minute
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 42
mean count per minute
  Week 26 | 19.74 (131.622)
  Week 52: number analyzed (Participants) | 20
  Week 52 | 44.58 (153.196)
  Week 78: number analyzed (Participants) | 10
  Week 78 | 99.14 (165.965)
  Week 104: number analyzed (Participants) | 2
  Week 104 | -62.87 (189.264)

ADVERSE EVENTS:
Time Frame: Up to 133 weeks
Description: The RUBATO open-label extension set (OLES) included all participants who were enrolled in this study and received at least 1 dose of macitentan 10 milligrams (mg).
Arm/Group | Macitentan 10 mg
All-Cause Mortality (participants affected / at risk) | 1/111
Serious Adverse Events (participants affected / at risk) | 18/111
Other Adverse Events (participants affected / at risk) | 34/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=111)
Arrhythmia (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Hepatic Mass (Hepatobiliary disorders) | 1
Covid-19 (Infections and infestations) | 1
Cytomegalovirus Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1
Sperm Concentration Decreased (Investigations) | 1
Spermatozoa Progressive Motility Decreased (Investigations) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Clonic Convulsion (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 — This data was not corresponding to a study participant but the female partner of a male participant.
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental Disorder (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=111)
Palpitations (Cardiac disorders) | 7
Fatigue (General disorders) | 7
Pyrexia (General disorders) | 3
Covid-19 (Infections and infestations) | 13
Pharyngitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5

LIMITATIONS AND CAVEATS:
The study was stopped prematurely by the sponsor because the main double-blind (DB) study (AC-055H301; NCT03153137) did not meet the primary and secondary efficacy outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 30 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03775421/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT03775421/SAP_002.pdf